CLINICAL TRIAL: NCT06519305
Title: Examination of Musculoskeletal System Problems, Pain and Quality of Life Related to Working Conditions in Chiropractors
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, AYCAN ÇAKMAK REYHAN, PhD, Istanbul Bilgi University
Other Study IDs: IstanbulBuu
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Problems, Pain, and QoL in Chiropractors in Relation to Their Working Conditions
Keywords: musculoskeletal system problems,; pain,; quality of life,; chiropractors
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey completion — Participants will be asked to fill out the survey via email.

SUMMARY:
This research aims to investigate musculoskeletal problems and pain, as well as their effects on the quality of life, arising from the working conditions of chiropractors in their workplaces. Additionally, it is intended to conduct a detailed analysis of working conditions in chiropractors' work environments to identify existing problems, establish the cause-and-effect relationship between musculoskeletal problems, pain, and these conditions, conduct studies to improve chiropractors' work environments, and demonstrate the positive effects of improving working conditions on the quality of life and professional performance of chiropractors. Within this scope, the physical layout of chiropractors' work environments, ergonomic factors, and workplace conditions will be analyzed. Musculoskeletal problems experienced by chiropractors will be identified, and research will be conducted on pain and musculoskeletal disorders associated with workplace factors. Furthermore, the effects of working conditions on the quality of life of chiropractors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female physiotherapists between the ages of 25-45, with at least 1 year of chiropractic experience, will be selected

Exclusion Criteria:

* Having practiced chiropractic for less than 1 year.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Professionals actively working as chiropractors
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | 1 mount
  VAS is a measurement tool commonly used to assess subjective characteristics or experiences, particularly pain intensity. It typically consists of a straight line, usually 10 centimeters in length, with one end representing the extreme of the characteristic being measured (e.g., "no pain" or "worst pain imaginable") and the other end representing the opposite extreme. Participants are asked to mark on the line the point that best represents their experience. This mark's distance from the zero point (e.g., "no pain") is then measured to quantify the characteristic being assessed. For pain intensity, the distance marked by the participant correlates with the severity of their pain, with longer distances indicating more severe pain. The VAS is a simple yet effective tool for quantifying subjective experiences and is widely used in clinical settings and research studies to assess various factors such as pain intensity, mood, and well-being.
SF-36 Short Form 36 Health Survey, | 1 mount
  The SF-36, or Short Form 36, is a widely used questionnaire designed to assess an individual's health-related quality of life. It consists of 36 questions that cover eight different health domains: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Each domain is scored separately, and the scores can be aggregated to produce two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). These summary measures provide an overall assessment of physical and mental health status, respectively. The SF-36 is a valuable tool in clinical research and healthcare settings for evaluating patients' overall health status, tracking changes over time, and comparing different patient populations.

SECONDARY OUTCOMES:
The Beck Depression Inventory (BDI) | 1 mount
  BDI), also known as the Beck Depression Scale, is a self-report questionnaire designed to measure the severity of depression symptoms in individuals. Beck, the BDI consists of 21 items that assess various symptoms commonly associated with depression, such as sadness, guilt, fatigue, changes in appetite or sleep patterns, and suicidal thoughts.Each item on the scale presents a statement describing a particular symptom, and individuals are asked to rate how much they have been experiencing each symptom over a specific time frame, typically the past two weeks. Responses are scored on a scale ranging from 0 to 3, with higher scores indicating greater severity of depressive symptoms.The total score on the BDI provides an overall measure of depression severity, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)